CLINICAL TRIAL: NCT04926480
Title: Comparison of the Effects of Low Flow and High Flow Anesthesia on Thiol-Disulfide Homeostasis and Ischemia Modified Albumin in Laparoscopic Cholecystectomy Surgery
Brief Title: Low Flow and High Flow Anesthesia on Thiol-Disulfide Homeostasis and IMA in Laparoscopic Cholecystectomy Surgery
Acronym: İMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, sermın emınoglu, specialist MD, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2011-KAEK-25 2019 /12-21
Record Dates: First submitted 2021-04-21; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Low Flow; High Flow; tiyol-disülfid homeostasis; Modified Albumin

STUDY DESIGN:
Masking Description: low flow high flow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low flow Anesthesia group (Experimental): Antioxidant parameters are measured in the low flow anesthesia group.
  Interventions: Procedure: low and high flow Anesthesia
- high flow Anesthesia gruop (Active Comparator): Antioxidant parameters are measured in the high flow anesthesia group.
  Interventions: Procedure: low and high flow Anesthesia

INTERVENTIONS:
Procedure: low and high flow Anesthesia — comparison of hemodynamic changes in low and high flow anesthesia groups
  Other Names: Cholecystectomy Surgery

SUMMARY:
Comparison of the Effects of Low Flow and High Flow Anesthesia on Thiol-Disulfide Homeostasis and Ischemia Modified Albumin in Laparoscopic Cholecystectomy Surgery

In this study, our aim is to compare the effects of Low Flow and High Flow Anesthesia on Thiol-Disulfide Homeostasis and Ischemia Modified Albumin in laparoscopic Cholecystectomy Surgery using Sevoflurane as an anesthetic gas routinely.

DETAILED DESCRIPTION:
General anesthesia is characterized by reversible loss of consciousness, analgesia in the whole body, amnesia, and some muscle relaxation. Induction, which is the initial phase of anesthesia, can be performed with intravenous or inhalation anesthetics. The most common practice today for maintenance of anesthesia after induction is to add an effective low intensity inhalation anesthetic to the oxygen, nitrous oxide or oxygen,air mixture. Although new inhalation agents provide some advantages over old ones, they are more costly. This situation has brought the development of new anesthetic techniques to the agenda. Interest in low fresh gas flow anesthesia methods has been increasing in recent years. The high standard of anesthesia machines, the availability of monitors that continuously analyze the anesthetic gas composition, and the increase in knowledge on the pharmacokinetics and pharmacodynamics of inhalation anesthetics have greatly facilitated the safe application of low-flow anesthesia. The term low flow anesthesia is used to describe inhalation anesthesia techniques with a semi closed rebreathing system with a reventilation rate of at least 50%, and with the help of a reversible anesthesia system, after the carbon dioxide is removed from the expired gas mixture from the patient, the metabolic requirements of the body are determined. At least 50% of the fresh oxygen flow is given back to the patient together with the volatile anesthetics in sufficient quantity. Many different anesthesia applications with different fresh gas flow rates have been described. Very high flow > 4 L / min, High flow 2-4 L / min, Medium flow 1-2 L / min, Low flow 500-1000 mL / min, Minimal flow 250-500 mL / min, Metabolic flow <250 mL / min. Currents of 1 L / min and below enter the low flow anesthesia head. The low flow anesthesia we use routinely has many advantages for the patient. Increasing the respiration rate of the humidified and warmed exhaled gas is of great importance for the function of the ciliated epithelium and for mucociliary cleaning, it provides a significant reduction in postoperative sore throat. It has an economic advantage due to the reduction in anesthetic gas consumption. It reduces exposure to anesthetic gases in the operating room environmen ; hypoxia, incompatibility of anesthesia depth, hypercarbia, possibility of heat accumulation and increased risk of bacterial contamination. Safety Features in Anesthesia Machines; According to the European common standard EN 740 conditions; They have features for monitoring inspired oxygen concentration, Monitoring of inhaled CO2 concentration, Monitoring of Volatile anesthetic concentration, Oxygen support insufficiency alarm, Oxygen bypass, Oxygen rate monitor. Although the risk is very low in low flow, oxygen in inspired fresh gas to avoid hypoxia Its concentration should be at least 50%. Depth of anesthesia can be adjusted according to the sevoflurane gas concentration in the monitor. Inspired and expired CO2 monitoring is important for patient safety. In order to prevent hypercarbia, appropriate carbon dioxide absorbent should be used and frequent replacement should be provided. Bacterial filters should also be used in the breathing circuit to prevent heat build-up and bacterial contamination. In high-flow anesthesia, drying of the respiratory tract and a decrease in mucociliary activity occurs. The use of a breathing circuit with a moisture retaining chamber and a moisture retaining filter can prevent this situation. Increasing anesthetic gas consumption increases the cost of the anesthetic gas in the surgical environment.

The use of volatile anesthetics such as desflurane or sevoflurane during general anesthesia causes an increase in lipid peroxidation or proinflammatory cytokines in macrophages, leading to generalized inflammatory reactions. It is stated that all these can cause oxidative stress, and under general anesthesia, patients are exposed to oxidative stress caused by volatile anesthetics. However, laparoscopic cholecystectomy, which has become a common procedure due to its advantages, increases the intraabdominal pressure, liver, splanchnic vessels, mesenteric hypoxia, ischemia. It causes reperfusion damage and consequently an increase in oxidative stress. Sevoflurane is a widely used anesthetic agent, its anti-inflammatory and antioxidant properties have been demonstrated in various studies, it has been shown that it protects against ischemia-reperfusion damage in vital organs such as heart, lung and kidney, and has more protective effects on thiol disulfide homeostasis than desflurane.

Thiols are compounds containing sulfur group, which are essential antioxidant buffers that interact with almost all physiological oxidants. Thiol groups are oxidized by the surrounding oxidant molecules and converted to disulfide structures and then thiol groups, thiol disulfide balance was a sustainable reaction. Thiols act as fast electron acceptors and play an important role in defending against reactive oxygen species by contributing a large part of the total antioxidants present in the body. Plasma thiols have pro-oxidant or antioxidant effects on physiological events; but they are generally regarded as antioxidants. It also plays a critical role in programmed cell death, detoxification, antioxidant protection and regulation of cellular enzymatic activity. Measuring thiols in serum may show an indirect reflection of antioxidant defense. Another oxidation parameter that can be used as a perioperative ischemia marker is ischemia-modified albumin (IMA). Hypoxia, acidosis, and superoxide radical damage cause IMA formation by altering the structure of the N terminal, reducing the binding capacity of albumin to metals. IMA is an early-rising indicator of ischemia, it increases in as little as 6 minutes. Anesthesia method, surgical method, medications used, infection and operation time affect postoperative morbidity and mortality by changing the stress response.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Aged 18-70 years
* elective laparoscopic cholecystectomy surgery
* general anesthesia

Exclusion Criteria:

* Morbidly obese patients
* alcohol or drug addiction
* chronic obstructive pulmonary disease
* coronary artery disease
* congestive heart failure
* significant anemia
* liver or kidney disease
* allergy to propofol or halogenated drugs
* respiratory system pathology, hypotension
* hypovolemia and patients with a systemic disease
* patients using drugs that may affect the oxidation system
* patients who are converted to open surgery intraoperatively and develop complications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the Effects of Low Flow and High Flow Anesthesia on Thiol-Disulfide Homeostasis and Ischemia Modified Albumin in Laparoscopic Cholecystectomy Surgery | 24 hours after operation
  In order to determine thiol / disulphid homeostasis and IMA serum level, 5 ml blood samples were taken 3 times from each patient (T0: 5 minutes before induction of anesthesia, T1: 5 minutes after abdominal gas is completely evacuated, T2: 24 hours postoperatively). Serum disulfide/thiol homeostasis measurements were determined by the automated spectrophotometric method described by Erel and Neşelioğlu.Thiol/disuphide hemostasis parameters were studied with the same serum samples in the same session. Ischemia modified albumen Bar-Or et al. The study was carried out using the spectrophotometric method suggested by The IMA is specified as the absorption unit (AUC).
Comparison of the Effects of Low Flow and High Flow Anesthesia on Thiol-Disulfide | during peroperative period
  During the operation, heart rate beats/min were recorded on the monitor at the 5th, 10th, 15th, 30th, 45th, 60th, 90th, 120th, 150th, 180th and 210th minutes after intubation and at the end of extubation.

CONTACTS AND LOCATIONS:
Overall Officials: umran karaca, 3, Study Director — Assistant researcher; asıye demirel, 4, Principal Investigator — Assistant researcher; mehmet gamlı, 5, Principal Investigator — Assistant researcher; yasemin ustundag, 6, Principal Investigator — Assistant researcher; ozcan erel, 7, Principal Investigator — Assistant researcher
Locations (2):
- Turkey (Türkiye) (2):
  - Bursa yüksek ihtisas training and research hospital, Bursa
  - Bursa yüksek ihtisas, Bursa

IPD SHARING:
Plan to Share IPD: No
Study protocol and results can be shared